CLINICAL TRIAL: NCT06227468
Title: A Clinical Study to Map the HLA GENomic Region and Its potEntial aSsocIation With Selected diSeases in the Greek Population
Brief Title: A Clinical Study to Map the HLA Genomic Region in the Greek Population
Acronym: GENESIS
Status: Recruiting | Type: Observational
Sponsor: Athens LifeTech Park (Other)
Collaborators: Galatea.Bio (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALTP.2023.001
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Respiratory Disease; Chronic Renal Failure; Cardiovascular Diseases; Metabolic Disease; Psychiatric Disorder; Neurologic Disorder; Gastrointestinal Diseases; Haematologic Disease; Rheumatologic Disease
MeSH Terms: conditions — Respiration Disorders; Kidney Failure, Chronic; Cardiovascular Diseases; Metabolic Diseases; Mental Disorders; Nervous System Diseases; Gastrointestinal Diseases; Hematologic Diseases; Collagen Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two buccal swabs per subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Greek population: The enrolled subjects will be managed as a single group.

SUMMARY:
The aim of GENESIS clinical study is to map the HLA genomic region in the Greek population and evaluate possible correlations with selected underlying diseases.

DETAILED DESCRIPTION:
The GENESIS study is a multicenter, prospective, non-interventional, clinical study with a target of 12,000 subjects and an anticipated total duration of 36 months. The aim of study GENESIS is to provide a pilot map of HLA genetic variation in the Greek population in order to be used in medical research and for possible clinical applications (evaluation of possible correlations with selected underlying diseases). During the study, each subject will conduct one visit to the participating cite, in which they will provide:

1. Demographic information [i.e. date of birth, gender, race, ancestry (including information about the subject's grandparents' birthplace), height, weight],
2. Other information about smoking/vaping, alcohol consumption, arterial blood pressure, diagnosed diseases (if any), current treatments (if any), and
3. Recent (up to 12 months prior to sample collection) results if/when are available from clinical lab tests such as blood count (Hct, Hb, RBC, WBC, PLT count), including a metabolic panel, liver enzymes and biochemical parameters (Glu, HbA1c, TC, TG, LDL-C, HDL-C, ALT, AST, ALP, γGT, bilirubin, LDH, insulin, C-peptide).

Upon completion of the data registry, two buccal swabs will be collected per subject and they will be stored at ALTP premises until their shipment to Galatea.Bio. All buccal swab samples will be subjected to genetic material (DNA) extraction. The DNA samples will be further proceeded for HLA genotyping analysis. A follow up analysis will be performed in selected DNA samples via full low-pass whole genome sequencing (LP-WGS), which aims to further investigate the association between the HLA region and autoimmune diseases.

Upon completion of the analysis, an individualized ancestry report will be securely made available to all study subjects which they can access, as and if they elect to.

ELIGIBILITY:
Inclusion Criteria:

The study will include adult subjects (age ≥ 18) that:

* possess a Greek social security number and are visiting hospitals/clinics, and/or other private laboratory institutions (incl. clinics and health care groups) as part of standard clinical practice in Greece,
* are willing and able to provide written informed consent to participate in the study according to the study protocol.

Exclusion Criteria:

* Subjects not able to provide written informed consent (e.g. ICU patients, mental illness patients, lack of legal capacity).
* Subjects who have had an allogeneic (non-self-donor):

  * bone marrow transplant
  * stem cell transplant
  * blood transfusion less than two weeks prior to buccal swab sample collection
  * liver transplant
* Subjects who participated in an interventional clinical trial in the past that according to the subject's physician opinion might have had an impact on their HLA genome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit and enroll eligible subjects possessing a Greek social security number, who are visiting hospitals/clinics and/or other private laboratory practices (incl. clinics and health care groups) as part of standard clinical practice.
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Allele frequency of HLA-alleles at the Greek population level | 36th month
  To assess the HLA allelic diversity of Greek population

SECONDARY OUTCOMES:
Prevalence of selected HLA-related diseases in the Greek population | 36th month
  Characterization of the allelic and haplotypic HLA frequency distribution in the Greek population and comparison with global HLA databases.
Relative Risk (Risk Ratio (RR) or Odds Ratio (OR)) of HLA markers on diseases of interest | 36th month
  Evaluation of the association between HLA alleles and/or haplotypes, and selected diseases

CONTACTS AND LOCATIONS:
Overall Officials: Efi Giannopoulou, Study Director — Athens LifeTech Park
Locations (8):
- Greece (8):
  - 2nd Propaedeutic Department of Internal Medicine, Attikon University General Hospital, Chaïdári, Attica
  - 2nd Department of Neurology, AHEPA University Hospital, Thessaloniki, Thessaloniki
  - Department of Respiratory Medicine, University General Hospital of Alexandroupolis, Alexandroupoli, Thrace
  - Department of Infectious Diseases, 2nd Department of Internal Medicine, University General Hospital of Alexandroupolis, Alexandroupoli
  - Department of Cardiology, University General Hospital of Heraklion, Heraklion
  - Department of Rheumatology, University Hospital of Heraklion, Heraklion
  - Department of Respiratory, University Hospital of Ioannina, Ioannina
  - Department of Haematology, University General Hospital of Larissa, Larissa

IPD SHARING:
Plan to Share IPD: No
No plan for sharing IPD at this stage

REFERENCES:
- [Background] Sanchez-Mazas A, Nunes JM, Middleton D, Sauter J, Buhler S, McCabe A, Hofmann J, Baier DM, Schmidt AH, Nicoloso G, Andreani M, Grubic Z, Tiercy JM, Fleischhauer K. Common and well-documented HLA alleles over all of Europe and within European sub-regions: A catalogue from the European Federation for Immunogenetics. HLA. 2017 Feb;89(2):104-113. doi: 10.1111/tan.12956. PMID 28102034
- [Background] Dendrou CA, Petersen J, Rossjohn J, Fugger L. HLA variation and disease. Nat Rev Immunol. 2018 May;18(5):325-339. doi: 10.1038/nri.2017.143. Epub 2018 Jan 2. PMID 29292391
- [Background] Zhou Y, Krebs K, Milani L, Lauschke VM. Global Frequencies of Clinically Important HLA Alleles and Their Implications For the Cost-Effectiveness of Preemptive Pharmacogenetic Testing. Clin Pharmacol Ther. 2021 Jan;109(1):160-174. doi: 10.1002/cpt.1944. Epub 2020 Jul 26. PMID 32535895